CLINICAL TRIAL: NCT06170372
Title: The Effectiveness of Adding Multiple Intermittent High-dose Inhalations of Nitric Oxide to Standard Antibacterial Therapy in the Treatment of Pneumonia
Brief Title: High-dose Inhalations of Nitric Oxide in the Treatment of Pneumonia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Principal Investigator, Tatiana P. Kalashnikova, MD, PhD, senior researcher of Laboratory, Tomsk National Research Medical Center of the Russian Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NO PNEUMONIA
Record Dates: First submitted 2023-12-06; First posted 2023-12-14 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Nosocomial Pneumonia; Community-acquired Pneumonia
MeSH Terms: conditions — Healthcare-Associated Pneumonia; Community-Acquired Pneumonia | interventions — Nitric Oxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Main group with nosocomial pneumonia (Experimental): Standard antibacterial therapy + Nitric Oxide 200 ppm 3 times a day for 30 minutes under the control of methemoglobin level (no more than 5%). The general course of Nitric Oxide therapy will last until the pneumonia resolves, but no more than 7 days.
  Interventions: Drug: 200 ppm Nitric Oxide
- Control group with nosocomial pneumonia (Active Comparator): Standard antibacterial therapy + medical air without Nitric Oxide 3 times a day for 30 minutes until the pneumonia resolves, but no more than 7 days.
  Interventions: Drug: Sham treatment
- Main group with community acquired pneumonia (Experimental): Standard antibacterial therapy + Nitric Oxide 200 ppm 3 times a day for 30 minutes under the control of methemoglobin level (no more than 5%). The general course of Nitric Oxide therapy will last until the pneumonia resolves, but no more than 7 days.
  Interventions: Drug: 200 ppm Nitric Oxide
- Control group with community acquired pneumonia (Active Comparator): Standard antibacterial therapy + medical air without Nitric Oxide 3 times a day for 30 minutes until the pneumonia resolves, but no more than 7 days.
  Interventions: Drug: Sham treatment

INTERVENTIONS:
Drug: 200 ppm Nitric Oxide — NO will be supplemented at 200-ppm concentration 3 times a day for 30 min until the pneumonia resolves, but no more than 7 days
  Other Names: nitrogen monoxide
  Arms: Main group with community acquired pneumonia; Main group with nosocomial pneumonia
Drug: Sham treatment — Oxygen-air mixture without NO 3 times a day for 30 min until the pneumonia resolves, but no more than 7 days
  Other Names: Oxygen-Air Mixture
  Arms: Control group with community acquired pneumonia; Control group with nosocomial pneumonia

SUMMARY:
This is a multicenter, prospective randomized controlled trial. At least 2 but no more than 5 centers are expected to participate in the study.

The primary objective is to test the hypothesis that the addition of high-dose inhaled nitric oxide therapy to standard treatment has a positive effect on the clinical course of pneumonia and the structure and function of cardiopulmonary system.

Number of participants: 200, including the subproject NO-PNEUMONIA-CAP - 100 CAP participants, the subproject NO-PNEUMONIA-NP - 100 NP participants.

Number of groups: 4 Inhalation of iNO at a dose of 200 ppm for 30 minutes under the control of methemoglobin level (no more than 5%) three times a day if the patient is allocated to the main group. The general course of iNO therapy will last until the pneumonia resolves, but no more than 7 days. Recording of vital signs and safety assessment will be carried out immediately before the initiation of NO therapy and every 15 minutes after its start (pulse, blood pressure, respiratory rate, SpO2, temperature, MetHb level).

DETAILED DESCRIPTION:
Principal investigator: T.P. Kalashnikova, MD, PhD. Sub-investigators: N.O.Kamenshchikov, MD, PhD, I.V. Kravchenko, MD, Yu.A. Arsenyeva, MD, Yu.K. Podoksenov, MD, PhD, DMedSci, M.S. Kozulin, MD, M.B. Gorchakova, MD, B.N. Kozlov, MD, PhD, DMedSci, A.A. Boshchenko, MD, PhD, DMedSci.

RESEARCH RELEVANCE Pneumonia remains one of the most common infectious respiratory diseases worldwide. Community-acquired pneumonia (CAP) is defined as pneumonia that is acquired outside the hospital or diagnosed in the first 48 hours from hospitalization. Nosocomial pneumonia (NP) is diagnosed in individuals with symptoms of the disease that develop 48 hours or more after the patient's hospitalization. The most common causative agents of CAP are S. pneumoniae, M. pneumoniae, C. pneumoniae, H. influenza, as well as viruses and microbial associations. In recent years, there has been an increase in the resistance of CAP pathogens to antibiotics of the group of aminopenicillins, cephalosporins, and macrolides.

In the etiological structure of NP, the leading role belongs to gram-negative microorganisms. The main pathogens are representatives of Enterobacteriaceae (including Klebsiella pneumoniae and E.coli), Acinetobacter baumannii, Pseudomonas aeruginosa, characterized by a high level of resistance to antimicrobial drugs.

Considering the high prevalence of pneumonia, the continuous increase in the resistance of microorganisms to antimicrobial agents, the high mortality rate from adverse reactions caused by multidrug-resistant bacteria, the lack of development of new drugs with proven antibacterial effectiveness, and the high economic costs of treatment, it is urgent to search for alternative ways to increase efficiency in the treatment of pneumonia . From this point of view, the addition of inhaled high doses of nitric oxide (iNO) to standard antibacterial therapy seems promising.

The positive results of using NO have been proven in the treatment of patients with pulmonary hypertension, chronic obstructive pulmonary disease, acute respiratory distress syndrome (ARDS), and in the treatment of wound processes. There is a cardioprotective and nephroprotective effect of this molecule that has been described. In recent years, data have appeared on the successful use of iNO in the treatment of viral pneumonia, in particular in pneumonia caused by the Severe acute respiratory syndrome-related coronavirus 2 (SARS-CoV2). High concentrations of nitric oxide cause cytotoxic, antibacterial, antiviral, and antifungal effects.

The use of iNO for pneumonia is pathogenetically justified. It has a selective vasodilating effect on pulmonary blood vessels with no systemic effect on hemodynamics. By reducing vascular resistance in the ventilated areas of lungs, it improves ventilation-perfusion ratio and can increase systemic oxygenation, reduce pulmonary hypertension and right ventricular dysfunction, and promotes the inclusion of previously unventilated alveoli in gas exchange.

The use of NO appears even more justified in the treatment of pneumonia in patients undergoing cardiac surgery under cardiopulmonary bypass (CPB), since their lungs are subject to ischemia and reperfusion injury during CPB.

In recent years, more and more evidence has emerged that the mechanisms of antimicrobial action of NO differ from those of modern traditional antibiotics, which is most relevant in the treatment of infections caused by multidrug-resistant bacteria and polymicrobial infections.

The antibacterial effect of NO at a dose of 160 ppm (parts per million) and higher has been described for a number of microorganisms. The safety of using iNO for humans in doses of 160-200 ppm for 15-30 minutes 2 to 5 times a day has been demonstrated in a number of clinical studies with Mycobacterium abscessus, other complex clinical situations, in patients with cystic fibrosis, in pregnant women and newborns. In contrast to bacterial membranes sensitive to NO, the stability of membranes of epithelial cells and fibroblasts and the absence of cytolysis when exposed to nitric oxide 200 ppm 3 times a day was proven in experimental studies and on cells of living human tissues.

PRIMARY OBJECTIVE To test the hypothesis that the addition of high-dose inhaled nitric oxide therapy to standard treatment has a positive effect on the clinical course of pneumonia and the structure and function of cardiopulmonary system.

SECONDARY OBJECTIVES

* To assess the timing of resolution of pneumonia in the main (with iNO) and control (without iNO) groups
* To assess differences in the dynamics of acute phase reactants in the main and control groups.
* To assess differences in the X-ray of the lungs and its dynamics in the main and control groups.
* To assess differences in variables of the functional state of the lungs and their dynamics according to spirometry and the 6-minute walk test under the influence of therapy in the main and control groups.
* To study differences in the dynamics of the main variables of the structural and functional state of the heart during echocardiography in the main and control groups.

The effectiveness of the study will be assessed by such a concept as "end point".

The primary composite endpoint will be resolution of pneumonia. The term "resolution of pneumonia" will include three criteria: achieving an oxygenation index SpO2/fraction of inspired oxygen (FiO2) >315; Respiratory Rate (RR)<20; discontinuation of antibacterial therapy.

Secondary hospital endpoints:

1. Difference in the duration of systemic inflammatory response syndrome (fever, leukocytosis, a shift in the white blood cells (WBC) towards more immature cells, increased levels of C-reactive protein (CRP), procalcitonin (PCT) in the study groups.
2. Difference in the duration of respiratory support in the study groups.
3. Difference in the frequency of changing antibacterial treatment regimens due to ineffectiveness in the compared study groups.
4. Difference in the frequency of transfer of patients to non-invasive ventilation (NIV), mechanical ventilation in the study groups.
5. Difference in the incidence of sepsis and septic shock in both groups.
6. Difference in the frequency of decrease in oxygen saturation after 72 hours from the start of therapy below 95% with an initially normal level or by 3% or more with an initially reduced level in the main and control groups.
7. Difference in the frequency of negative computer tomography (CT) dynamics after 72 hours of therapy in the study groups.
8. Difference in the frequency of increase in right atrial and ventricle volume index and/or peak tricuspid regurgitation velocity and/or decrease in contractile function of the right ventricle after 72 hours of therapy and with the resolution of pneumonia in groups
9. Difference in the distance traveled according to the 6-minute walk test (6MWT) with the resolution of pneumonia in the main and control groups.
10. Difference in the frequency and severity of the development of ventilatory disorders during spirometry at the time of resolution of pneumonia in the main and control groups.
11. Difference in scores according to EQ-5D-5L quality of life questionnaire in the main and control groups.
12. Difference in the percentage of mortality caused by pneumonia or its complications (sepsis, multiple organ failure, acute respiratory failure) in the compared groups.

The study will include patients who underwent cardiac surgery under CPB with NP diagnosed in the postoperative period, as well as patients hospitalized for CAP. Patients will be randomized into 4 groups:

Subproject NO-PNEUMONIA-NP Group 1, main group, n=50 Standard antibacterial therapy + NO 200 ppm 3 times a day for 30 minutes Group 2, control group, n=50, Standard antibacterial therapy Subproject NO-PNEUMONIA-CAP Group 3, main group, n=50 Standard antibacterial therapy + NO 200 ppm 3 times a day for 30 minutes Group 4, control group, n=50 Standard antibacterial therapy. A special device, which synthesizes nitric oxide from atmospheric air directly during therapy, will be used. The technology is based on the process of oxidation of atmospheric nitrogen in a nonequilibrium gas discharge plasma and is characterized by high operating accuracy and stable maintenance of NO concentration in the breathing mixture.

ASSESSMENT OF CLINICAL EFFECTIVENESS Clinical effectiveness will be assessed daily with registration of data at control points (day of development of pneumonia, 72 hours from the onset of the disease, resolution of pneumonia) according to the dynamics of the temperature curve, oxygen saturation (SpO2), respiratory rate, oxygenation index SpO2∕FiO2, assessment of quality of life according to European Quality-of-Life-5 Dimension (EQ -5D-5L) questionnaire.

LABORATORY ASSESSMENT Laboratory effectiveness will be assessed by the levels of peripheral blood leukocytes, the significance of blood shift in the leukocyte formula, the dynamics of CRP, PCT (screening, 72 hours from the onset of the disease, resolution of pneumonia).

ASSESSMENT OF INSTRUMENTAL EFFICIENCY

1. Distance traveled during the 6-minute walk test on the day the pneumonia resolved.
2. Spirometry will be performed on the day of screening and on the day of resolution of pneumonia and include assessment of Vital capacity, Forced vital capacity, Forced expiratory volume in one second, Peak expiratory flow, Forced expiratory flow at 25% of Forced vital capacity (FVC), Forced expiratory flow at 50% of FVC, Forced expiratory flow at 75% of FVC.
3. Chest CT scan on the day of screening, after 72 hours and on the day of resolution of pneumonia with determination of localization and size of consolidation, localization and size of the Ground-glass opacity, air bronchograms (yes/no), hemodynamic abnormalities (yes/no), fluid volume in the pleural cavities.
4. Cardiac ultrasound will be performed on the day of screening, 72 hours later, and on the day of resolution of pneumonia and will include assessment of end-diastolic, end-systolic volume indexes and left ventricular ejection fraction, right ventricular antero-posterior diameter, right ventricular fractional area change, tricuspid regurgitation velocity, Tricuspid annular plane systolic excursion (TAPSE) , tricuspid annular systolic velocity (S'), right ventricular free wall longitudinal strain (if possible), diameter of the inferior vena cava and its collapse during inspiration, fluid in the pericardial cavity (yes/no, volume insignificant/moderate/severe/tamponade ) and pleural cavities.

ELIGIBILITY:
Inclusion Criteria:

1. An established diagnosis of Nosocomial Pneumonia (NP) after cardiac surgery under cardiopulmonary bypass (CPB) or hospitalization for Community-acquired pneumonia (CAP).
2. Spontaneous breathing.
3. Age > 18 years.
4. Signed informed consent.
5. Negative result of immunochromatographic Severe acute respiratory syndrome-related coronavirus 2 rapid antigen test on the day of diagnosis of pneumonia.

Diagnostic criteria for NP The diagnosis of NP is considered established when the number of points on the

Clinical Pulmonary Infection Score (CPIS) is greater than 6:

Diagnostic criteria for CAP:

Radiologically confirmed focal pulmonary opacity and at least 2 clinical symptoms and signs of the following:

1. acute fever at the onset of the disease (t° > 38.0°C);
2. cough with sputum;
3. physical signs (crepitus/fine rales, bronchial breathing, shortening of percussion sound);
4. leukocytosis > 10x109/l and/or left shift (> 10%)

Exclusion Criteria:

1. Diagnosed infectious process of another localization (surgical site infection (SSI), acute and chronic urinary tract infection (active), catheter-related bloodstream infection, peritonitis, infective endocarditis etc.).
2. Mechanical ventilation
3. Presence of tracheostomy
4. Patient's participation in another clinical trial at the time of screening or within the previous 3 months.
5. Concomitant pulmonary disease with the need for respiratory support before the development of pneumonia.
6. History of malignancy or other irreversible diseases/conditions with a life expectancy of less than 1 year.
7. Presence of HIV infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Pneumonia resolution time (days) | 30 days from the date of randomization
  Pneumonia resolution time is assessed as number of days from the date of randomization till pneumonia resolution.

SECONDARY OUTCOMES:
Fever higher than 37˚C (days) | 30 days from the date of randomization
  Fever is assessed in number of days when the level of fever is higher than 37˚C
Total leukocyte counts (10*9/L) | 72 hours from the start of therapy
  The difference in the levels of leukocytes (counts) is assessed between the time points corresponding to the start of therapy and 72 hours after therapy begins in the study groups
Immature cell counts (percentage) | 72 hours from the start of therapy
  The difference between the levels of immature cells (counts) in the leukocyte formula is assessed between the time points corresponding to the start of therapy and 72 hours after therapy begins in the study groups
Pneumonia resolution-associated change in total leukocyte counts (10*9/L) | 30 days from the date of randomization
  The difference in the levels of leukocytes (counts) is assessed between the time points corresponding to the start of therapy and the day of pneumonia resolution. In case pneumonia does not resolve within 30 days, the change is assessed between the date of randomization and day 30.
Pneumonia resolution-associated change in immature cell counts (percentage) | 30 days from the date of randomization
  The difference in the levels of leukocytes (counts) is assessed between the time points corresponding to the start of therapy and the day of pneumonia resolution. In case pneumonia does not resolves within 30 days, the change is assessed between the date of randomization and day 30.
C-reactive protein (CRP) level | 72 hours from the start of therapy
  The difference in the levels of C-reactive protein (mg/L) is assessed between the time points corresponding to the start of therapy and 72 hours after therapy begins.
Pneumonia resolution-associated change in C-reactive protein level (mg/L) | 30 days from the date of randomization
  The difference in the levels of C-reactive protein (mg/L) is assessed between the time points corresponding to the start of therapy and the day of pneumonia resolution. In case pneumonia does not resolves within 30 days, the change is assessed between the date of randomization and day 30.
Procalcitonin (PCT) level (ng/mL) | 72 hours from the start of therapy
  The difference in the levels of procalcitonin (PCT) (ng/mL) is assessed between the time points corresponding to the start of therapy and 72 hours after therapy begins.
Pneumonia resolution-associated change in procalcitonin (PCT) level (ng/mL) | 30 days from the date of randomization
  The difference in the levels of procalcitonin (PCT) (ng/mL) is assessed between the time points corresponding to the start of therapy and the day of pneumonia resolution. In case pneumonia does not resolves within 30 days, the change is assessed between the date of randomization and day 30.
Respiratory support time (days) | 30 days from the date of randomization
  Respiratory support time is assessed as number of days when respiratory support is required.
Frequency of changing antibacterial treatment regimens (times) | 30 days from the date of randomization
  Frequency of changing antibacterial treatment regimens is assessed as number of modifications to antibacterial treatment required due to its ineffectiveness.
Incidence of sepsis (percentage) | 30 days from the date of randomization
  Incidence of sepsis is assessed as percentage of cases.
Incidence of septic shock (percentage) | 30 days from the date of randomization
  Incidence of septic shock is assessed as percentage of cases.
Incidence of oxygen saturation decrease (percentage) | 30 days from the date of randomization
  Incidence of oxygen saturation decrease is assessed as percentage of cases where patients with initially normal oxygen saturation level have oxygen saturation below 95% and/or patients with initially reduced oxygen saturation level have a drop in oxygen saturation by 3% and more after 72 hours the start of therapy.
Incidence of adverse computer tomography (CT) findings (percentage) | 72 hours from the start of therapy
  Incidence of adverse computer tomography (CT) findings is assessed as percentage of cases with adverse findings on CT on day 3 after the start of therapy.hours of therapy in the study groups
Right atrial volume index (RAVI) (mL/m2) | 72 hours from the start of therapy
  Right atrial volume index (RAVI) (mL/m2) is measured by echocardiography at day 3 after the start of therapy
Right ventricular volume index (mL/m2) | 72 hours from the start of therapy
  Right ventricular volume index (RAVI) (mL/m2) is measured by echocardiography at day 3 after the start of therapy.
Pneumonia resolution-associated right atrial volume index (RAVI) (mL/m2) | 30 days from the date of randomization
  Right atrial volume index (RAVI) (mL/m2) is measured by echocardiography on the day of pneumonia resolution.
Pneumonia resolution-associated right ventricular volume index (mL/m2) | 30 days from the date of randomization
  Right ventricular volume index (mL/m2) is measured by echocardiography on the day of pneumonia resolution.
Increased peak tricuspid regurgitation velocity (percentage) | 72 hours from the start of therapy
  Incidence of increase in peak tricuspid regurgitation velocity is assessed as percentage of cases on day 3 after the start of therapy.
Increased peak tricuspid regurgitation velocity (percentage) | 30 days from the date of randomization
  Incidence of increase in peak tricuspid regurgitation velocity is assessed as percentage of cases on day 30 after the start of therapy.
Six-minute walk test (6MWT) distance (meters) | 30 days from the date of randomization
  Six-minute walk test (6MWT) distance (meters) is assessed at the day of pneumonia resolution. In case pneumonia does not resolves within 30 days, the 6MWT distance is assessed on day 30.
Lung vital capacity (L) | 30 days from the date of randomization
  Lung vital capacity is assessed in liters (L) at the day of pneumonia resolution. In case pneumonia does not resolve within 30 days, lung vital capacity is assessed at day 30.
Forced vital capacity (L) | 30 days from the date of randomization
  Forced vital capacity is assessed in liters (L) at the day of pneumonia resolution. In case pneumonia does not resolve within 30 days, forced vital capacity is assessed on day 30.
Forced expiratory volume (L/s) | 30 days from the date of randomization
  Forced expiratory volume is assessed in liters per second (L/s) at the day of pneumonia resolution. In case pneumonia does not resolve within 30 days, forced expiratory volume is assessed on day 30.
Peak expiratory flow (L/s) | 30 days from the date of randomization
  Peak expiratory flow is assessed in liters per second (L/s) at the day of pneumonia resolution. In case pneumonia does not resolve within 30 days, peak expiratory flow is assessed on day 30.
Quality of life (score) | 72 hours from the date of randomization
  Quality of life is assessed according to EQ-5D-5L quality of life questionnaire score on day 3 after the start of therapy.
Quality of life (score) | 30 days from the date of randomization
  Quality of life is assessed according to EQ-5D-5L quality of life questionnaire score at the day of pneumonia resolution. In case pneumonia does not resolve within 30 days, quality of life is assessed on day 30
Mortality caused by pneumonia or its complications (percentage) | 30 days from the date of randomization
  Mortality due to pneumonia or its complications is assessed as percentage

CONTACTS AND LOCATIONS:
Overall Officials: Tatiana P Kalashnikova, MD, PhD, Principal Investigator — Cardiology Research Institute, Tomsk National Research Medical Center
Locations (1):
- Cardiology Research Institute Tomsk National Research Medical Center, Tomsk, Select..., Russia